CLINICAL TRIAL: NCT03092440
Title: Validity Assessment of the "LabForGames Warning" Serious Game
Status: Completed | Type: Observational
Sponsor: Université Paris-Sud (Other)
Responsible Party: Principal Investigator, Antonia Blanie, Antonia Blanie M D, Université Paris-Sud
Other Study IDs: LabForSIMS-002
Record Dates: First submitted 2017-03-14; First posted 2017-03-28 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Education
Keywords: Medical Education; simulation; serious game; validity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- "Nursing students" group: nursing students
  Interventions: Other: serious game
- "New nurses" group: Nurses with < 2 years experience
  Interventions: Other: serious game
- "Expert nurses" group: Intensive nurses (with ≥ 4 years experience post graduate)
  Interventions: Other: serious game

INTERVENTIONS:
Other: serious game — During three hours, each learner will play with the three different cases of the "LabForGames Warning" serious game.

SUMMARY:
The use of simulation in medical education has been associated with positive results in the acquisition of knowledge, skills, behaviors and patient outcome. Serious games are useful educational tools since they allow both theory and practice training for an important number of learners, simultaneously. However, few studies have evaluated the validity and effectiveness of serious games.

Our simulation unit (LabForSIMS- Faculté de Médecine Paris-Sud, France) has developed a serious game named "LabForGames Warning" for nursing students with the following learning objectives: to recognize and to address the degradation of a patient's clinical condition and to work on the issue of inter-professional communication. The aim of the present study is to determine content and construct validities of the "LabForGames Warning" serious game before its use as a healthcare professional training tool.

DETAILED DESCRIPTION:
This observational single-center open study will be conducted in the simulation center of the Paris-Sud medical school (LabForSIMS). After written consent, the study population (nurses and nursing students) will attend a three hours simulation session with the "LabForGames Warning" serious game and will be divided into three groups :

* Nursing students
* New Nurses: Nurses with < 2 years experience
* Expert Nurses: Intensive nurses, with ≥ 4 years experience post graduate.

During three hours, each learner will play with the three different cases of the "LabForGames Warning" serious game then an auto-evaluation will be recorded.

The primary outcome measure was the evaluation of the construct validity:

The score (/100) and the duration (min) of each case of the serious game will be reported in order to assess whether the difference of the measures is related to the difference of skills between the three groups. An auto-evaluation of clinical reasoning will also be recorded.

The secondary outcome measure was the evaluation of content and face validities. For content validity, the content and parameters will be tested by the nurses ≥ 4 years experienced (Ten-point Likert scale) For face validity, the students' satisfaction and the resemblance between the virtual game and the real life clinical practice will be evaluated in the three groups (Ten-point Likert scale).

ELIGIBILITY:
Inclusion Criteria:

* Nursing students or nurses with < 2 years experience or intensive nurses (with ≥ 4 years experience post graduate)
* and having agreed to participate

Exclusion Criteria:

* Subjects incapable of giving consent: incapacitated (subjects under guardianship), minors (< 18 years)
* Refusal to participate in to the study Refusal to sign in the confidentiality clause

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Voluntary divided into three groups :
  * "Nursing students" group
  * "New nurses" group: Nurses with < 2 years experience
  * "Expert nurses" group: Intensive nurses (with ≥ 4 years experience post graduate)
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
The score (/100) of each case of the serious game | 60 min
  The score (/100) of each case of the serious game will be reported in order to assess whether the difference of the measures is related to the difference of skills between the three groups (Evaluation of the construct validity). An auto-evaluation of clinical reasoning will also be recorded.
the duration (min) of each case of the serious game | 60 min
  The duration (min) of each case of the serious game will be reported in order to assess whether the difference of the measures is related to the difference of skills between the three groups (Evaluation of the construct validity).

SECONDARY OUTCOMES:
The content and parameters of the serious game | 30 min
  For content validity, the content and parameters of the serious game will be tested by the nurses ≥ 4 years experienced (Ten-point Likert scale)
Learners' satisfaction | 5 min
  For face validity, the learners' satisfaction and the resemblance between the virtual game and the real life clinical practice will be evaluated in the three groups (Ten-point Likert scale).
The resemblance between the virtual game and the real life clinical practice | 25 min
  For content validity, the resemblance between the virtual game and the real life clinical practice will be evaluated in the three groups (Ten-point Likert scale).

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Blanié, M.D, Principal Investigator — Université Paris Sud, 91 400 Orsay, France
Locations (1):
- Faculté de médecine Paris Sud, Le Kremlin-Bicêtre, France

REFERENCES:
- [Derived] Blanie A, Amorim MA, Meffert A, Perrot C, Dondelli L, Benhamou D. Assessing validity evidence for a serious game dedicated to patient clinical deterioration and communication. Adv Simul (Lond). 2020 May 27;5:4. doi: 10.1186/s41077-020-00123-3. eCollection 2020. PMID 32514382